CLINICAL TRIAL: NCT02839824
Title: Evaluation of the Quality of Bowel Cleansing in a Real Clinical Practice Setting (CALICOL Study)
Brief Title: Evaluation of the Quality of Bowel Cleansing in a Real Clinical Practice Setting
Acronym: CALICOL
Status: Completed | Type: Observational
Sponsor: Casen Recordati S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAS-EVA-2016-01
Record Dates: First submitted 2016-07-14; First posted 2016-07-21 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: bowel cleansing; bowel preparation
MeSH Terms: interventions — Cathartics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Bowel preparation — Bowel preparation for bowel cleansing in a real clinical practice

SUMMARY:
Publications of the use of bowel cleansers in usual clinical practice are lacking. Patient adherence to investigational products increases in the context of clinical trials. By the same token, efficacy of interventions may be overestimated in clinical trials.

For this reason, an observational study to collect data on the effectiveness of several colonic preparations when these are used under usual clinical practice is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Subjects who have been performed a colonoscopy

Exclusion Criteria:

* Subjects being previously performed colon surgery.
* Subjects suffering from active inflammatory bowel disease at the time of performing colonoscopy.
* Subjects with extreme limitations due to disease.
* Subjects in who Boston Bowel Preparation Scale (BBPS) is not available
* Subjects who have undergone a colonoscopy during their participation in another clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have been performed a colonoscopy and who have received a bowel cleansing agent according to the investigator criteria
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with adequate colon cleansing | Through study completion, an average of 6 months
  Percentage of patients with punctuation in Boston bowel preparation scale (BBPS) ≥ 5

SECONDARY OUTCOMES:
Percentage of patients with adequate colon cleansing of different administration schedules | Through study completion, an average of 6 months
  Percentage of patients with punctuation in BBPS ≥ 5 in each administration schedule
Identify factors influencing bowel cleansing quality | Through study completion, an average of 6 months
  Relationship between BBPS ≥ 5 and age, gender, ethnicity, weight, height, tobacco consumption, concomitant diseases, medications and indication for colonoscopy in a multivariate analysis.
Influence of total volume of liquid ingestion in the effectiveness of bowel cleansing agents | Through study completion, an average of 6 months
  Relationship between BBPS ≥ 5and the volume of liquid ingestion
Patients' tolerance | Through study completion, an average of 6 months
  Percentage of each adverse event reported per patient in each administration schedule
Quality of bowel cleansing comparison among different bowel cleansing agents | Through study completion, an average of 6 months
  Comparison of percentage of patients with BBPS ≥ 5 between different bowel cleansing agents
Subjects' satisfaction | Through study completion, an average of 6 months
  Comparison of subjects' satisfaction between different bowel cleansing agents with a five point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Ana Bargalló, MD, Study Director — Clínica de Medicina Integral Diagonal, Gastroenterology department
Locations (1):
- Clínica de Medicina Integral Diagonal, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No